CLINICAL TRIAL: NCT04166110
Title: A Controlled Randomized, Open Label, Multicenter, Non-inferiority Trial Evaluating an Individualized Antibiotic Duration Treatment Based on Patient Clinical Response, Evaluated Through Connected Devices, for Community Acquired Pneumonia in the Community Setting
Brief Title: Antibiotic Therapy In Respiratory Tract Infections
Acronym: AIR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P160929J; 2019-001873-10 (EudraCT Number)
Record Dates: First submitted 2019-09-30; First posted 2019-11-18 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Community-Acquired Pneumonia
Keywords: community-acquired pneumonia; antibiotic therapy duration strategy; non-inferiority trial
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physician's prescription (Active Comparator): Antibiotic treatment duration according to physician, following the French national guidelines: 7 to 14 days.
  Interventions: Drug: Predetermined treatment duration
- Duration according to stability (Experimental): Antibiotic treatment duration is variable. Interruption of treatment is based on the patient reaching stability criteria (body temperature ≤ 37.8°C; heart rate ≤ 100/min; systolic blood pressure ≥ 90mmHg, oxygen saturation ≥ 90%).
  Minimum of duration of antibiotic treatment: 3 days.
  Interventions: Drug: Variable treatment duration

INTERVENTIONS:
Drug: Predetermined treatment duration — Antibiotic treatment duration left to the physician's judgement (following national guidelines, 7 to 14 days)
  Arms: Physician's prescription
Drug: Variable treatment duration — Treatment duration vary according to stability criteria reaching time Patients will self-monitor 2 times a day (in the morning and in the evening) using a set of connected devices, to monitor their vital signs before any treatment intake.
  After at least 3 days of treatment and stability criteria obtained for the last 24 hours (i.e. 3 vital signs recording), patients will stop the antibiotic treatment.
  Arms: Duration according to stability

SUMMARY:
Primary aim: to demonstrate that stopping antibiotic treatment in patients diagnosed with acute community acquired pneumonia (CAP) based on clinical response has a non-inferior efficacy 15 days after start of treatment, compared to a conventional predetermined duration left to the physician's judgement, in adults treated in the community setting.

Secondary aims: To compare the 2 study arms on:

1. Clinical success at late follow up (Day 30),
2. Duration of antibiotic treatment,
3. Frequency and severity of adverse events,
4. Patient's pneumonia symptoms and quality of life.

DETAILED DESCRIPTION:
Recent studies have suggested that CAP can be successfully treated by short-course antibiotic regimen when clinical improvement is rapidly obtained. Even if clinical response is obtained in 3 days in the majority of cases, it can widely vary among patients, suggesting that "one duration does not fit all". An individualized duration of therapy depending on the patient's response could help to ensure bacterial eradication while avoiding unnecessary antibiotic exposure and thus reduce antibiotic resistance. At present, this strategy has never been tested.

This is a pragmatic open label non-inferiority randomized multicenter trial with two parallel arms comparing antibiotic treatment duration left to the physician's judgement (usually 7 to 14 days), versus interruption of treatment based on the patient's clinical response defined by reaching stability criteria (body temperature ≤ 37.8°C; heart rate ≤ 100/min; systolic blood pressure ≥ 90mmHg, oxygen saturation ≥ 90%) for 24h, after a minimum of 2 days treatment.

Recruitment and follow-up: Outpatients consulting in a private multiprofessional health center, diagnosed as having CAP and in need for antibiotics will be assessed for eligibility. Following information and signing consent, eligible patients will be included in the study. They will receive the prescription (antibiotic type and duration determined by the physician, preferably chosen according to the French guidelines) and a collection of connected devices to monitor their vital signs 2 times a day (morning and evening). Preselected patients will be randomized as soon as they meet the two following criteria: i) they have presented the stability criteria for 24h (3 consecutive vital signs recordings); ii) they have started the antibiotic treatment at least 72 hours before, with a ≥ 80% compliance, and with at least 1 intake in the last 24 hours. Each patient will then receive a telephone call from the coordinating team (or a permanent medical platform at nights, during weekends or public holidays) in order to proceed to the randomization and ensure that everything is well understood by the patient as well as the security and compliance with the strategy.

A follow-up visit with the investigator will be performed at day 15 after the start of antibiotic treatment.

The final evaluation will be performed 30 days following the start of antibiotic treatment by a telephone call from the coordinating team.

Number of subjects necessary: 310 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or more
* Has given written informed consent
* Affiliated to Health insurance
* Is able to take oral treatment
* Presenting with suspected CAP defined by the presence of at least 2 of the following diagnostic clinical criteria:

  * Fever (temperature > 38°C)
  * Dyspnea
  * Cough
  * Production of purulent sputum
  * Crackles
  * Radiological evidence of a new infiltrate (on chest X-ray or CT scan)
* In need for antibiotic treatment targeting respiratory tract, according to the physician in charge
* No other site of infection besides respiratory

Exclusion Criteria:

All subjects meeting any of the following exclusion criteria at baseline will be excluded from study participation:

* Signs of severe CAP (abscess, massive pleural effusion, serious chronic respiratory insufficiency)
* Hospitalization following consultation
* Known immunosuppression (asplenia, neutropenia, agammaglobulinemia, immunosuppressive treatments or corticosteroids (prednisolone equivalent) > 10 mg/day, transplant, myeloma, lymphoma, known HIV and CD4<400/mm3, sickle-cell disease, Child-Pugh class C cirrhosis)
* Suspected or confirmed legionellosis
* Atrial fibrillation / constitutive tachycardia
* Baseline oxygen saturation < 90% or home oxygen therapy
* More than 24 hours of antibiotics prior to consultation
* Any other infection necessitating concomitant antibiotic treatment
* Contraindications to the study antibiotics
* Concomitant steroid treatment only for patients treated with fluoroquinolones antibiotics
* Pre-existing aortic aneurysm or dissection, family history of aortic aneurysm or dissection, Marfan syndrome, Ehlers-Danlos syndrome, Takayasu arthritis, arterial hypertension, atherosclerosis only for patients treated with fluoroquinolones antibiotics
* Pregnancy
* Breastfeeding
* Life expectancy < 1 month
* Patient under legal guardianship or without healthcare coverage
* Homeless patient
* Patient enrolled in another interventional clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cure rate at day 15 | Day 15
  Cure rate is the number of patients who are cured, as defined by the association of 3 criteria :
  1. stability: body temperature ≤ 37.8°C; heart rate ≤ 100/min; systolic blood pressure > 90mmHg and oxygen saturation ≥ 90%.
  2. absence of: incidence of coughing, sputum production, shortness of breath and crackles.
  3. absence of additional antibiotic taken after the end of initial antibiotic treatment.
  Clinical evaluation at Day 14 or Day 16 is allowed to take into account.

SECONDARY OUTCOMES:
Cure rate at day 30 | Day 30
  Cure rate is the number of patients who are cured, as defined by the association of 2 criteria:
  1. absence of: incidence of coughing, sputum production, shortness of breath and crackles.
  2. absence of additional antibiotic taken after the end of initial antibiotic treatment.
Duration of antibiotic treatment | Up to 14 days
Frequency and severity of adverse events | through study completion, an average of 30 days
Evolution of pneumonia symptoms | through study completion, an average of 30 days
  Patients' evolution of pneumonia symptoms and quality of life between the 2 study arms (CAP Score / CAP Sym)

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien DINH, MD, Principal Investigator — Unité des Maladies Infectieuses, Hôpital Raymond Poincaré, Garches; Anne-Claude CRÉMIEUX, MD, PhD, Study Director — Service des maladies infectieuses, Hôpital Saint Louis, Paris
Locations (1):
- Unité des Maladies Infectieuses, CHU Raymond Poincaré, Garches, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No